CLINICAL TRIAL: NCT04535804
Title: Clinical Randomized Controlled Trial of Aspirin in the Treatment of Pregnant Women With Adenomyosis on Reducing Preterm Delivery
Brief Title: Aspirin in the Treatment of Pregnant Women With Adenomyosis on Reducing Preterm Delivery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KS20253
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Adenomyosis of Uterus
MeSH Terms: conditions — Adenomyosis | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin group (Active Comparator): 100 mg of low-dose aspirin was given orally (2 tablets a time, twice a day, before going to bed) to 36 weeks of gestation.
  Interventions: Drug: Aspirin/placebo
- placebo group (Placebo Comparator): 100 mg of placebo was given orally (2 tablets a time, twice a day, before going to bed) to 36 weeks of gestation.
  Interventions: Drug: Aspirin/placebo

INTERVENTIONS:
Drug: Aspirin/placebo — By using a random, double-blind research method, 1-550 digital computers are randomly divided into two groups, with two groups of digital coding placebo and aspirin. From 12 weeks of gestation, 100 mg of placebo or low-dose aspirin was given orally (2 tablets a time, twice a day, before going to bed) to 36 weeks of gestation.
  Other Names: acetylsalicylic acid

SUMMARY:
Objective: This study intends to carry out a randomized double-blind clinical trial study of aspirin in the treatment of pregnancy with adenomyosis to reduce the incidence of preterm delivery, and provide a new therapeutic target for the prevention and treatment of premature birth and adverse pregnancy outcomes, and fill in the blank of effective prevention of premature delivery in pregnancy with adenomyosis at home and abroad Application value and social and economic benefits of the bed.

Methods: a randomized double-blind clinical trial was used in this study. In Shanghai first maternal and child health care hospital, the pregnant women who meet the requirements of the group will be given full informed consent. By using a random, double-blind research method, 1-550 digital computers are randomly divided into two groups, with two groups of digital coding placebo and aspirin. From 12 weeks of gestation, 100 mg of placebo or low-dose aspirin was given orally (2 tablets a time, twice a day, before going to bed) to 36 weeks of gestation.

Observe the outcome ① Main outcome measures: preterm delivery: delivery less than 37 weeks gestational weeks, premature delivery. The specific classification includes: A. extremely premature delivery, gestational age 28-32 weeks; B. early preterm birth, delivery gestational weeks 32-34 gestational weeks; C. late preterm birth, 34-36 gestational weeks.

② Secondary outcome measures: abortion, gestational diabetes mellitus, gestational hypertension, placental disorders, SGA / FGR, premature rupture of membranes, postpartum hemorrhage, mode of delivery, etc.

The follow-up contents were as follows

* Routine prenatal examination, blood pressure, fetal size, vaginal bleeding, etc.

  * Coagulation factor index: prothrombin time Pt, activated partial thrombin time APTT, thrombin time TT, fibrinogen FIB, D-dimer

    * Immune related indexes: antiphospholipid antibody, CA125 ④ Inflammatory index: routine blood test + CRP

      * Detection of cervical length by B-ultrasound ⑥ Pregnancy complications: gestational diabetes mellitus, gestational hypertension and placental disorders ⑦ Birth outcome: gestational weeks, birth weight, FGR, premature delivery, mode of delivery, NICU rate, etc.

DETAILED DESCRIPTION:
Research background:

Adenomyosis (AD) is a benign uterine disease with endometrial glands and stroma invading into the myometrium, accompanied by hyperplasia and hypertrophy of uterine smooth muscle cells, which leads to abnormal uterine structure and function. In non pregnancy period, the main manifestations are diffuse enlargement of uterus, dysmenorrhea, menorrhagia, menorrhagia, which can lead to infertility. In recent years, with the delay of childbearing age, the incidence of adenomyosis in pregnancy is increasing gradually. The incidence of adenomyosis in the general population reached 20.9%, while the incidence of adenomyosis was higher in recurrent abortion and assisted reproduction, reaching 38.2% and 34.7% respectively. Studies have shown that adenomyosis is associated with early preterm delivery, late preterm delivery, low birth weight infants, very low birth weight infants, and small for gestational age infants. Patients with adenomyosis are prone to hypertensive disorder complicating pregnancy, intrauterine infection, abnormal placenta, and increased cesarean section, postpartum hemorrhage and abnormal fetal position.

Aspirin is widely used in the treatment of immune system diseases and the prevention of cerebrovascular diseases because of its anti-inflammatory and anti platelet aggregation effects. Aspirin is more and more widely used in obstetrics and Gynecology, such as recurrent abortion caused by antiphospholipid antibody syndrome, recurrent abortion related to abnormal uterine artery blood flow and unexplained recurrent abortion. Since 1980, aspirin has been widely recommended for the prevention of pregnancy with high risk factors of preeclampsia and intrauterine growth restriction, and it has been confirmed that aspirin is effective in the prevention of pregnancy It is safe in clinical application. The inflammatory environment of adenomyosis is closely related to the initiation of preterm delivery, but whether aspirin can benefit pregnant women with adenomyosis is still lacking.

Research plan

1. Study population Inclusive criteria: ① Singleton; ② in line with the diagnosis of adenomyosis in pregnancy; ③ no history of chronic diseases and definite diagnosis of endocrine diseases, including diabetes, hypertension, obesity, antiphospholipid syndrome; ④ informed consent and voluntary participation in this study.

   Exclusion criteria: ① twins / multiple births; ② induced labor for medical reasons; ③ allergic to aspirin or other salicylates, tetracycline drugs or any other components of drugs; ④ patients with mental disorders; ⑤ transferred to hospital.

   Withdrawal criteria: Subjects withdraw informed consent; subjects request to withdraw from the trial.

   Termination of the experiment: unacceptable adverse events occurred; the subjects voluntarily asked to withdraw from the trial; the protocol was violated; the researcher / ethics committee considered it necessary for the subjects to stop the trial.
2. Diagnostic criteria of adenomyosis: according to pre pregnancy and early pregnancy transvaginal ultrasound diagnosis. The diagnostic criteria of transvaginal ultrasound for adenomyosis include: (a) ectopic endometrial glands and stroma, (b) myometrium hyperplasia, hypertrophy, and increased blood vessels.
3. Sample size calculation: the incidence of preterm delivery in pregnant women with adenomyosis was about 21.63% (Mette R. Bruun et al. 2018). It is expected that the incidence of preterm birth in patients with adenomyosis during pregnancy will be reduced by 40% after aspirin intervention, that is, the incidence of premature delivery in the intervention group will be about 12.98%. Assuming that the test level α is 0.05, the test efficiency is 0.8, and one-sided test, 236 sample sizes are estimated for the intervention group and the control group by using the sample size estimation software pass. Considering the loss of follow-up rate of about 10%, the sample size of intervention group and control group was about 262 cases. Therefore, 550 pregnant women were recruited in this study.
4. Statistical analysis plan: the statistical analysis in the study is based on the principle of intention to treat (ITT), that is, all the subjects involved in the study participate in the statistical analysis. Chi square test or unpaired t test was used to analyze the difference between the intervention group and the control group. In the chi square test, if the theoretical frequency of cells was less than 5, Fisher exact probability method was used, and the Mann Whitney U test was used for quantitative variables that did not conform to normal distribution. Chi square test was used to analyze the difference of preterm birth rate between intervention group and control group. Logistic regression model was used to estimate the relative risk value and 95% confidence interval (95% confidence interval) of preterm birth between the two groups. The choice of statistical analysis method for secondary outcome indicators was consistent with that in primary outcome analysis. SAS viya was used as the analysis software in the study, and the difference was statistically significant when p < 0.05.

research implementation process: research steps (describe the data collection content and method according to the time node) 2020.10-2020.12：we distributed recruitment advertisements, prepared placebos and aspirin, screened and enrolled patients, signed informed consent, and arranged outpatient follow-up of enrolled patients; 2021.01-2021.06：150 cases of pregnant women with adenomyosis were planned to be enrolled, and the registration and follow-up of the patients were done well; 2021.07-2021.12：150 cases of pregnant women with adenomyosis were planned to be enrolled; the experimental data were summarized gradually; the information of defect was recorded; 2022.01-2022.06：150 cases of pregnancy with adenomyosis were planned to be enrolled, the pregnancy outcomes of the pregnant women were counted, and the case report forms were completed; 2022.07-2022.09： we plan to complete the work of 50 cases of pregnancy with adenomyosis, analyze the data statistically, write papers and final reports.

Risk of study: placebo had no effect on subjects; adverse reactions of aspirin mainly included gastrointestinal reactions, risk of fetal teratogenesis before 12 weeks of pregnancy, and risk of bleeding during pregnancy. However, since 1980, aspirin has been widely used in the prevention of pregnancy with high risk factors of preeclampsia and fetal growth restriction, which proves that the probability of adverse reactions of low-dose aspirin is very low, no teratogenic effect is found, and it has clinical safety.

Benefits of the study: expected to reduce the incidence of preterm birth and improve adverse pregnancy outcomes. In order to explore the prevention and treatment of premature delivery and adverse pregnancy outcomes, it is necessary to provide a new therapeutic target, fill in the blank of the effective prevention of premature birth treatment of pregnancy combined with adenomyosis at home and abroad, which may reduce the medical costs related to pregnancy complications and adverse pregnancy outcomes, as well as the cost of dealing with adverse pregnancy outcomes. This study has important clinical application value and social and economic benefits.

Recruitment and protection measures of subjects There are recruitment advertisements in this study, and other documents are provided; Protective measures for the subjects: in order to reduce the adverse reactions of aspirin as far as possible, we used aspirin enteric coated tablets, 50mg, twice a day, the dosage belongs to low dose. From 12 weeks of gestation to 36 weeks of gestation. If you have bleeding during pregnancy, you need to stop taking aspirin, and you can continue to take aspirin after the bleeding disappears. The number of follow-up visits during pregnancy is roughly the same as that of general prenatal examination (about 10 times), without additional visits; about 5ml more blood will be drawn for examination on the day of establishing pregnancy card, and the extra examination cost will be borne by the research group; we will arrange experienced doctors to take charge of the whole pregnancy examination of the subjects and keep communication at any time. We will pay more attention to the subject's gastrointestinal reaction, tinnitus, erythema, liver and kidney function and other discomfort during each birth examination. If there is any abnormality, we will take the following measures: (1) immediately stop your experiment if the condition requires; (2) be responsible for the treatment of your adverse drug reactions; (3) give appropriate economic compensation according to the degree of your injury.

Informed consent process: the subject's informed consent work is in charge of a specially assigned person, who will provide sufficient and easy to understand information to the pregnant women who meet the inclusion conditions; the subjects of informed consent are all those with independent ability, and they will not be able to participate in this project if they have no independent ability; there will be no pressure on pregnant women who meet the inclusion conditions in the process of informed consent. In the process of participating in the research, it will ensure that research participants get timely information (including their rights, safety and health).

ELIGIBILITY:
Inclusion Criteria:

* ① Singleton; ② in line with the diagnosis of adenomyosis in pregnancy; ③ no history of chronic diseases and definite diagnosis of endocrine diseases, including diabetes, hypertension, obesity, antiphospholipid syndrome; ④ informed consent and voluntary participation in this study.

Exclusion Criteria:

* ① twins / multiple births; ② induced labor for medical reasons; ③ allergic to aspirin or other salicylates, tetracycline drugs or any other components of drugs; ④ patients with mental disorders; ⑤ transferred to hospital.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 550 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
preterm delivery | Gestation 12-36 weeks
  delivery less than 37 weeks gestational weeks, premature delivery. The specific classification includes: A. extremely premature delivery, gestational age 28-32 weeks; B. early preterm birth, delivery gestational weeks 32-34 gestational weeks; C. late preterm birth, 34-36 gestational weeks.

SECONDARY OUTCOMES:
Other complications | Gestation 12-36 weeks
  abortion, gestational diabetes mellitus, gestational hypertension, placental disorders, SGA / FGR, premature rupture of membranes, postpartum hemorrhage, mode of delivery, etc.

CONTACTS AND LOCATIONS:
Overall Officials: qiaoling Du, doctorate, Study Chair — Shanghai first maternal and infant hospital

IPD SHARING:
Plan to Share IPD: No